CLINICAL TRIAL: NCT01797068
Title: Patient Navigation to Improve Care and Reduce Costs for High Utilizers of the Emergency Department
Brief Title: Patient Navigation for Medicaid Frequent ED Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1007007154
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2016-11

CONDITIONS: Chronic Illness
Keywords: HEALTHCARE UTILIZATION; ED UTILIZATION; PRIMARY CARE UTILIZATION; PATIENT NAVIGATION; UNDERSERVED POPULATIONS; HEALTH DISPARITIES
MeSH Terms: conditions — Chronic Disease | interventions — Patient Navigation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigator (Experimental): Patients in the experimental group will be offered patient navigation and timely access to comprehensive care and services through Project Access-New Haven (PA-NH).
  Interventions: Behavioral: Patient Navigator
- Standard of Care (Active Comparator): Patients in the active comparator group will experience the usual intake process in the ED setting.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Patient Navigator — Patients in the intervention group will be offered patient navigation and timely access to comprehensive care and services through Project Access-New Haven (PA-NH), a local non-profit organization that coordinates the provision of donated medical care and services to underserved patients through a network of participating hospitals and volunteer physicians.
  Arms: Patient Navigator
Other: Standard of Care — Patients in the standard of care group will experience the usual intake process in the ED setting.
  Arms: Standard of Care

SUMMARY:
A large proportion of frequent ED users have Medicaid insurance. The purpose of this study is to evaluate the effectiveness of patient navigation for reducing Emergency Department (ED) visits and hospitalizations and improving patient-centered outcomes (e.g., self-reported health status, quality of life, access/barriers to care) among Medicaid patients who are high utilizers of the ED, as well as to identify best practices for engaging and providing healthcare services to underserved patients using patient navigation. This study will address needs that have been identified within the New Haven community and the local healthcare system, contribute to knowledge and literature surrounding the use of patient navigation to improve care for underserved patients and improve health system efficiency, and inform the design and development of programs that address these needs both locally and in other communities.

ELIGIBILITY:
Inclusion Criteria:

* 4-18 ED visits per year
* Frequent ED users
* age 18 to 62
* Medicaid insurance only
* Those living in the greater New Haven area (i.e. having a zip code that matches that)

Exclusion Criteria:

* the current visit for primary psychiatric or substance abuse
* more than 50% of all ED visits in the past year for primary psychiatric or substance abuse.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of ED visits | One Year
  Additional outcomes include number of hospitalizations, number of outpatient visits, and outpatient imaging utilization.

SECONDARY OUTCOMES:
Number of hospitalizations | One Year
Number of outpatient visits | One Year
Costs by analyzing global use with Medicaid claims data | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States